CLINICAL TRIAL: NCT03499535
Title: Impact of Smoking Information on Concerns About Radon
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Paul Windschitl (Other)
Responsible Party: Sponsor-Investigator, Paul Windschitl, Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 201507727
Record Dates: First submitted 2018-03-30; First posted 2018-04-17 (Actual); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: Lung Neoplasms; Radon Exposure; Smoking; Intention; Risk Reduction Behavior
Keywords: Risk Perception
MeSH Terms: conditions — Lung Neoplasms; Smoking; Risk Reduction Behavior | interventions — Radon

STUDY DESIGN:
Intervention Model Description: Study 1: Participants randomly assigned to one of two conditions. Study 2: Participants randomly assigned to one of three conditions.
Who Masked: Participant
Masking Description: Participants blinded to condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Study 1: Radon&Smoking Synergistic/EPA (Active Comparator): Participants viewed radon and smoking risk information taken from the EPA's pamphlet on the dangers of radon gas exposure.
  Interventions: Behavioral: Radon & Smoking Synergistic; Behavioral: EPA
- Study 1: Radon&Smoking Synergistic/Idaho (Active Comparator): Participants viewed radon and smoking risk information taken from Idaho's Department of Health and Human Welfare's pamphlet on the dangers of radon gas exposure.
  Interventions: Behavioral: Radon & Smoking Synergistic; Behavioral: Idaho
- Study 1: Radon Only / EPA (Experimental): Participants viewed only radon risk information taken from the EPA's pamphlet on the dangers of radon gas exposure.
  Interventions: Behavioral: Radon Only; Behavioral: EPA
- Study 1: Radon Only / Idaho (Experimental): Participants viewed only radon risk information taken from Idaho's Department of Health and Human Welfare's pamphlet on the dangers of radon gas exposure.
  Interventions: Behavioral: Radon Only; Behavioral: Idaho
- Study 2: Radon Only (Experimental): Participants viewed a radon-only message that focused only on the effect of radon on lung-cancer risk.
  Interventions: Behavioral: Radon Only
- Study 2: Radon and Smoking Isolated (Other): Participants viewed a radon-and-smoking-isolated message that covered the individual effects of radon and of smoking on lung cancer, but without mentioning their synergistic effect.
  Interventions: Behavioral: Radon and Smoking Isolated
- Study 2: Radon & Smoking Synergistic (Active Comparator): Participants viewed a radon-and-smoking-synergistic message that covered the individual effects of radon and of smoking but that also included information about their synergistic effect.
  Interventions: Behavioral: Radon & Smoking Synergistic

INTERVENTIONS:
Behavioral: Radon & Smoking Synergistic — Participants viewed health information detailing the risks of developing lung cancer from exposure to radon gas, smoking, and their synergistic effects. This intervention represents the type of information most commonly presented in radon risk communications.
  Arms: Study 1: Radon&Smoking Synergistic/EPA; Study 1: Radon&Smoking Synergistic/Idaho; Study 2: Radon & Smoking Synergistic
Behavioral: Radon Only — Participants viewed health information detailing the risks of developing lung cancer from radon exposure. No information about the risks for developing lung cancer associated with smoking or its synergistic effect with radon exposure are included.
  Arms: Study 1: Radon Only / EPA; Study 1: Radon Only / Idaho; Study 2: Radon Only
Behavioral: Radon and Smoking Isolated — Participants viewed health information detailing the risks of developing lung cancer from radon exposure and smoking. No information describing the synergistic effects of smoking and radon exposure on lung cancer risk are included.
  Arms: Study 2: Radon and Smoking Isolated
Behavioral: EPA — Health information modeled after the Environmental Protection Agency's (EPA) pamphlet on radon risk.
  Arms: Study 1: Radon Only / EPA; Study 1: Radon&Smoking Synergistic/EPA
Behavioral: Idaho — Health information modeled after the Idaho Department of Health and Human Welfare's pamphlet on radon risk.
  Arms: Study 1: Radon Only / Idaho; Study 1: Radon&Smoking Synergistic/Idaho

SUMMARY:
Despite a push for tailored messages, health communications are often aimed at, and viewed by, people with varying levels of risk. This project examined-in the context of radon risk messages-whether information relevant to high-risk individuals can have an unintended influence on lower-risk individuals. Specifically, the investigators assessed whether information about lung-cancer risk from smoking reduced concerns about lung-cancer risk from radon among nonsmokers. The investigators hypothesized that non-smokers who read a message that included smoking-relevant information would express less concern about the effects of radon exposure and less interest in testing their home compared to those who read a version in which smoking-relevant information was excluded. Two studies were conducted. Although the investigators did not exclude smokers, the focus was on participants self-identifying as nonsmokers (including never smokers and former smokers).

DETAILED DESCRIPTION:
Despite a push for tailored messages, health communications are often aimed at, and viewed by, people with varying levels of risk. This project examined-in the context of radon risk messages-whether information relevant to high-risk individuals can have an unintended influence on lower-risk individuals. Specifically, the investigators assessed whether information about lung-cancer risk from smoking reduced concerns about lung-cancer risk from radon among nonsmokers. The investigators hypothesized that non-smokers who read a message that included smoking-relevant information would express less concern about the effects of radon exposure and less interest in testing their home compared to those who read a version in which smoking-relevant information was excluded. Two studies were conducted. Although the investigators did not exclude smokers, the focus was on participants self-identifying as nonsmokers (including never smokers and former smokers). Participants in both studies were recruited through Amazon's Mechanical Turk (MTurk). Participants viewed radon messages that varied in the information they communicated about smoking's effect on lung cancer. In Study 1, smoking information was included or excluded from messages assembled from existing radon pamphlets. In Study 2, versions of a new radon message either excluded smoking information, described smoking as a major cause of lung cancer, or also described smoking's synergistic effect with radon on lung cancer risk. After viewing a radon health message, participants completed a variety of measures. Primary measures assessed respondents' anticipated sense of concern and related reactions if they learned that they/their home had been exposed to elevated levels of radon. Other key measures included questions about participants' interest and intention to test their home for radon.

ELIGIBILITY:
Inclusion Criteria:

* Live within the US
* Have an Amazon Mechanical Turk account (website where online study was posted)

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1390 (Actual)
Dates: Start 2015-08-07 (Actual); Primary Completion 2016-04-22 (Actual); Study Completion 2016-04-22 (Actual)

PRIMARY OUTCOMES:
Conditional Concern Composite | Immediately post-intervention (approx. 1 minute)
  Composite formed from 4 conditional questions assessing concern, perceived impact on risk and comparative risk, and threat--if exposed to radon
Interest in Testing Composite | Immediately post-intervention (approx. 2 minutes)
  Composite formed from 2 questions assessing importance and intention to test home for radon

SECONDARY OUTCOMES:
Worry Elicited by Health Message | Immediately post-intervention (approx. 2 minutes)
  Single question assessing worry elicited by the health communication material
Likelihood Judgments about Lung Cancer | Immediately post-intervention (approx. 4 minutes)
  Three items assessing perceived likelihood of developing lung cancer
Elect to Leave Email for Raffle | Immediately post-intervention (approx. 4 minutes)
  Participants given option to leave email address in case they won one of the 20 radon kits being raffled (Study 2).
Elect to Read More | Immediately post-intervention (approx. 4 minutes)
  Participants given option to be presented with more information at the end of the session about testing for radon (Study 2).
Concern about Loved Ones If Exposed to Radon | Immediately post-intervention (approx. 4 minutes)
  Rated how concerned they would be about loved ones if they learned their home had high radon (Study 2)

IPD SHARING:
Plan to Share IPD: Yes
De-identified data and guide will be made available to other investigators upon request.
Supporting Information: Analytic Code
Time Frame: Requested data will be made available upon publication of the project.
Access Criteria: Please contact corresponding author Dr. Paul Windschitl at paul-windschitl@uiowa.edu